CLINICAL TRIAL: NCT05488405
Title: Open-label, Monocentric Phase IIa Pilot Study Evaluating the Efficacy and Tolerability of a 4-week Treatment With Mesalazine Oral Suspension in Patients With Active Eosinophilic Esophagitis
Brief Title: Mesalazine Oral Suspension in Active Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAV-1/EEA
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Eosinophilic Esophagitis
Keywords: Esophageal dysfunction, esophageal inflammation
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophageal Diseases; Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesalamine treatment (Experimental): Treatment of patient with mesalamine oral suspension
  Interventions: Drug: Mesalamine Oral Product

INTERVENTIONS:
Drug: Mesalamine Oral Product — Mesalamine oral suspension for oral use
  Other Names: 5-ASA

SUMMARY:
Pilot study to assess a mesalazine oral suspension in active eosinophilic esophagitis

DETAILED DESCRIPTION:
This is an open-label, monocentric exploratory phase IIa pilot study, which serves to evaluate the efficacy, safety, and tolerability of treatment with mesalazine oral suspension for the treatment of active eosinophilic esophagitis (EoE).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female patients, 18 to 75 years of age
* Confirmed clinico-pathological diagnosis of eosinophilic esophagitis (EoE) according to established diagnostic criteria
* Negative pregnancy test in females of childbearing potential

Exclusion Criteria:

* Other causes for esophageal eosinophilia
* Clinical and endoscopic signs of gastroesophageal reflux disease (GERD)
* Any concomitant esophageal disease and relevant gastro-intestinal disease (celiac disease, inflammatory bowel disease, oropharyngeal or esophageal bacterial, viral, or fungal infection [candida esophagitis])
* Any known or suspicion for relevant infectious diseases associated with clinical signs,
* Known intolerance/hypersensitivity/resistance to the IMP or excipients or drugs of similar chemical structure or pharmacological profile
* Existing or intended pregnancy or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with histological remission | 4 weeks
  Assessment of remission of histological signs of EoE

SECONDARY OUTCOMES:
Proportion of patients with histological response | 4 weeks
  Assessment of improvement of histological signs of EoE
Proportion of patients with improvement of symptoms | 4 weeks
  Clinical symptoms will be assessed via patient reported outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Biedermann, PD Dr. med., Principal Investigator — UniversitätsSpital Zürich Klinik für Gastroenterologie und Hepatologie
Locations (1):
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No